CLINICAL TRIAL: NCT02726477
Title: Efficacy and Safety of Wuling San on Breast Cancer-related Lymphedema
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fourth Affiliated Hospital of Guangxi Medical University (Other)
Collaborators: Liuzhou Maternity and Child Healthcare Hospital (Other); Liuzhou Hospital of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PJK2016088
Record Dates: First submitted 2016-03-29; First posted 2016-04-01 (Estimated); Last update posted 2016-05-09 (Estimated); Status verified 2016-05

CONDITIONS: Breast Cancer; Lymphedema
MeSH Terms: conditions — Breast Neoplasms; Lymphedema

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Wuling San (Experimental): This is a double-blinded, randomized placebo-controlled, multi-center clinic trial, using before and after treatment measurements.
  A total of 200 clinical diagnosed BCRL participants with affected arm circumference 10-40% larger than unaffected arm, are randomly allocated to two groups: the Wuling San group or the placebo group, where the intervention group administers Wuling San, at a dosage of 1g/kg, twice a day for six weeks. The primary outcome measurement will be the percentage of limb volume changes measured by perometry.
  Interventions: Drug: Wuling San
- placebo (Placebo Comparator): A total of 200 clinical diagnosed BCRL participants with affected arm circumference 10-40% larger than unaffected arm, are randomly allocated to two groups: the Wuling San group or the placebo group, where the placebo group administers a placebo powder, at a dosage of 1g/kg, twice a day for six weeks. The primary outcome measurement will be the percentage of limb volume changes measured by perometry.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Wuling San — Patients will be administrated with Wuling San at a dosage of 1g/kg twice a day after randomisation.
  Arms: Wuling San
Drug: placebo — Patients will be administrated with placebo powder at a dosage of 1g/kg twice a day after randomisation.
  Arms: placebo

SUMMARY:
The purpose of this study is to assess the efficacy and safety of Wuling San, a traditional Chinese medicine, in reducing arm volume excess in women with stage I-II breast cancer related unilateral lymphedema.

DETAILED DESCRIPTION:
The investigators will aim to enroll 200 female adult patients (aged between 20 and 40 years) of all ethnicities/races, who have been referred to the Fourth Affiliated Hospital of Guangxi Medical University for breast cancer related unilateral lymphedema. The investigators will be using a standardized data collection form in this study, where standard of care will be practiced and the patients are not placed at additional risk from participating in this study. However, as the investigators are collecting data prospectively, all participants will sign consent.

ELIGIBILITY:
Inclusion Criteria:

* Women completed all primary and adjuvant treatments (surgery, chemotherapy, radiotherapy)
* age 20-40 with unilateral BCRL, stage I or II, BMI of 18-25
* Volume difference ≥300 mL between the normal and lymphedematous upper extremity based on perometry evaluation
* No evidence of breast cancer recurrence
* At least 6 months postoperative from axillary lymph node dissection

Exclusion Criteria:

* Bilateral lymphedema or stage III lymphedema
* History of bilateral axillary lymph node dissection
* Recent history of cellulitis in the affected extremity (within last 3 months)
* Recurrent breast cancer or other malignancy
* Current (within last month) use of chemotherapy for breast or other malignancy
* Current (within last 3 months) use of radiation for breast or other malignancy
* Recent (within last month) or current intensive MLD and/or short stretch bandage use
* Unstable lymphedema (i.e. worsening symptoms/measurements in the past 3 months)
* Pregnant or nursing (lactating) women
* Patients that take drugs like diosmin at the time of enrollment, or within 30 days.
* Use of other investigational drugs at the time of enrollment, or within 30 days or 5 half-lives of enrollment, whichever is longer.
* Unable to comply with the protocol, measurement and follow-up schedule.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2016-04; Primary Completion 2017-09 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
volume changes % measured by perometry | baseline and 2 months
  Volume changes in the arm after the therapy will be calculated using the methods established by Anderson et al (2000). Briefly, the difference in volume measurements between the normal and lymphedematous arms at baseline will be compared to the volume differential after drug treatment (i.e volume excess) using the following formula:
  Change in absolute edema=(Vo-Vc)B-(Vo-Vc)3 months/(Vo-Vc)B
  Change in ln ratio=ln (Vo/Vc)B-ln (Vo/Vc)3 months.
  Vo is the volume of the lymphedema arm. Vc is the volume of the contralateral arm.
  Andersen, L., Højris, I., Erlandsen, M., & Andersen, J. (2000). Treatment of breast-cancer-related lymphedema with or without manual lymphatic drainage: a randomized study[J]. Acta Oncologica, 2000, 39(3): 399-405.

SECONDARY OUTCOMES:
adverse events | baseline and 2 months
  number of participants with serious and non-serious adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Xiangcheng Wei, Principal Investigator — Guangxi Medical University Institutional Review Board
Locations (3):
- China (3):
  - Liuzhou Hospital of Traditional Chinese Medicine, Liuchow, Guangxi
  - Liuzhou Maternity and Child Healthcare Hospital, Liuchow, Guangxi
  - The Fourth Affiliated Hospital of Guangxi Medical University, Liuchow, Guangxi

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Andersen L, Hojris I, Erlandsen M, Andersen J. Treatment of breast-cancer-related lymphedema with or without manual lymphatic drainage--a randomized study. Acta Oncol. 2000;39(3):399-405. doi: 10.1080/028418600750013186. PMID 10987238
- [Derived] Zhu H, Peng Z, Dai M, Zou Y, Qin F, Chen J, Song L, He B, Lv X, Dai S. Efficacy and safety of Wuling San for treatment of breast-cancer-related upper extremity lymphoedema: study protocol for a pilot trial. BMJ Open. 2016 Dec 16;6(12):e012515. doi: 10.1136/bmjopen-2016-012515. PMID 27986736